CLINICAL TRIAL: NCT04115774
Title: Registry of Osteogenesis Imperfecta That Collects Clinical, Functional, Genetic, Genealogical, Imaging, Surgical, Quality of Life Data. Data is Linked to Patients Biological Samples, When Available
Brief Title: Registry of Osteogenesis Imperfecta
Acronym: ROI
Status: Recruiting | Type: Observational
Sponsor: Luca Sangiorgi (Other)
Responsible Party: Sponsor-Investigator, Luca Sangiorgi, Head of Departement of Rare Skeletal Disorders, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: 21632/2013
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Osteogenesis Imperfecta
Keywords: Disease Registry; Natural History Study; Disease Evolution; Genotype-Phenotype Correlation
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Diphosphonates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — Whole peripheral blood, DNA, lymphocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteogenesis Imperfecta patients: The group comprises all patients affected by Osteogenesis Imperfecta, including prenatal and fetal diagnosis of Osteogenesis Imperfecta
  Interventions: Drug: bisphosphonates

INTERVENTIONS:
Drug: bisphosphonates — Since this is an observational study, the investigators collect general information on bisphosphonates treatment/impact

SUMMARY:
ROI is a retrospective and prospective registry, finalized for care and research purposes. It is articulated in main sections - strongly related and mutually dependent on each other - corresponding to different data domains: personal information, clinical data, genetic data, genealogical data, surgeries, etc. This approach has been developed to corroborate and integrate data from different sources evaluating several aspects of diseases and to correlate genetic background and phenotypic outcomes, in order to better investigate diseases pathophysiology. Due to legal requirements, institutional directives and organizational issues, we are unable to include individuals residing outside Italy in the registry at this time. We are currently engaged in the preparation of a recruitment process for individuals residing outside Italy.

DETAILED DESCRIPTION:
The traditional method of collecting patient information is often chaotic, inconvenient and sometimes even unsafe, particularly when dealing with rare diseases. In 2013, the need to simplify the diagnostic process and to overcome the difficulties of data storage and analysis, led to the suggestion of implementing the Registry of Osteogenesis Imperfecta (ROI).

The ROI relies on an IT platform named Genotype-phenotype Data Integration platform - GeDI. This solution was developed through a collaboration between Rare Skeletal Disease Department and a local software company (Dilaxia) and is General Data Protection Regulation (GDPR)-compliant, multi-client and web-accessible. It has been designed according to current medical informatics standards, including the Orphanet code, the International Classification of Diseases (ICD), the Human Genome Variants Society, aiming to follow FAIR (Findability Accessibility Interoperability Reusability) principles. GeDI is continuously being implemented to improve the management of people with Osteogenesis Imperfecta and to assist researchers in analyzing the information collected. ROI is divided into the following main sections:

* Personal data: it comprises general information, birth details and residence data;
* Patient data: including the patients internal code, the hospital code and other patient details;
* Diagnostic Process: the diagnosis, the status (affected, suspected, etc.), age at diagnosis, comorbidities, allergies, etc.;
* Genogram: a tool for designing the family transmission of the disease, alongside information on the disease status of all relatives included;
* Clinical events: it records a long list of signs and symptoms of Multiple Osteochondromas as well as several additional items to describe the disease
* Genetic Analysis and Alteration: including analytical technique, sample information, analysis duration, etc. This section also comprises detailed information on any detected pathological variants (e.g. gene, international reference, DNA change, protein change, genomic position, etc.);
* Visits: this section includes visit type (genetic, orthopedic, rehabilitation, pediatric, etc.), the date of the visit, prescriptions, imaging, etc.;
* Treatments: this section comprises information of a wide range of treatments including pharmacological, devices, supplements, and other treatments such as psychological, nutritional, etc.;
* Surgeries: this section contains information on the type of surgeries, the age of the patients, the site/localization of the procedures, etc.
* Documents: this repository allow us to store all types of documents (radiological reports, imaging, consents, clinical reports, etc.);
* Consents: this section provides a comprehensive overview of all consents collected, including the collection date;
* Samples: this section includes information on the samples, like the type, date of collection, etc.;
* PROs: this section collects information on patients reported outcomes such as the quality of life or ABC scale.

ELIGIBILITY:
Inclusion Criteria:

* All Osteogenesis Imperfecta patients, including prenatal and fetal diagnosis of Osteogenesis Imperfecta

Exclusion Criteria:

* Any condition unrelated to Osteogenesis Imperfecta

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by Osteogenesis Imperfecta. The Registry will include also data on foetuses (prenatal and abortion).
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-06-28 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2032-02-29 (Estimated)

PRIMARY OUTCOMES:
Natural History and Epidemiology | 25 years
  To maintain an established registry in order to assess epidemiology and natural history. Collection of physical examinations (severity of the disease), orthopaedics and functionals data (number of fractures, fracture sites, deafness, etc.), genetics background (target gene, type of mutation, etc.), family history (inheritance in maternal or paternal line, etc.) and treatment information (pharmacological, devices, supplements, and other treatments).
  Clinical, orthopedic, surgical, treatment and functional features are updated at each follow up. Clinical reports, medical charts and imaging are the primary source of data.

SECONDARY OUTCOMES:
Genotype-Phenotype Correlation | 25 years
  The secondary outcome comprises the correlation between genotype and phenotype. This includes, but is not limited to clinical features and genetic background. This will be pursued using the information collected during visits and follow-ups and the genetic information resulting from molecular investigations.

OTHER OUTCOMES:
Disease evolution | 25 years
  This outcome aims to investigate the evolution of Osteogenesis Imperfecta during time. This will be evaluated within the families and among the families.
  Main clinical features, such as height, number of fractures, bone evaluations, will be collected both retrospectively and prospectively. An evaluation of these parameters will be performed at each visit to keep track on the progression of clinical manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Sangiorgi, PhD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Ablin DS, Sane SM. Non-accidental injury: confusion with temporary brittle bone disease and mild osteogenesis imperfecta. Pediatr Radiol. 1997 Feb;27(2):111-3. doi: 10.1007/s002470050079. PMID 9028840
- [Background] Davie MW, Haddaway MJ. Bone mineral content and density in healthy subjects and in osteogenesis imperfecta. Arch Dis Child. 1994 Apr;70(4):331-4. doi: 10.1136/adc.70.4.331. PMID 8185368
- [Background] Chapman S, Hall CM. Non-accidental injury or brittle bones. Pediatr Radiol. 1997 Feb;27(2):106-10. doi: 10.1007/s002470050078. PMID 9028839
- [Background] Lindert U, Cabral WA, Ausavarat S, Tongkobpetch S, Ludin K, Barnes AM, Yeetong P, Weis M, Krabichler B, Srichomthong C, Makareeva EN, Janecke AR, Leikin S, Rothlisberger B, Rohrbach M, Kennerknecht I, Eyre DR, Suphapeetiporn K, Giunta C, Marini JC, Shotelersuk V. MBTPS2 mutations cause defective regulated intramembrane proteolysis in X-linked osteogenesis imperfecta. Nat Commun. 2016 Jul 6;7:11920. doi: 10.1038/ncomms11920. PMID 27380894
- [Background] Martin E, Shapiro JR. Osteogenesis imperfecta:epidemiology and pathophysiology. Curr Osteoporos Rep. 2007 Sep;5(3):91-7. doi: 10.1007/s11914-007-0023-z. PMID 17925189
- [Background] Miller ME, Hangartner TN. Temporary brittle bone disease: association with decreased fetal movement and osteopenia. Calcif Tissue Int. 1999 Feb;64(2):137-43. doi: 10.1007/s002239900592. PMID 9914321
- [Background] Moore MS, Minch CM, Kruse RW, Harcke HT, Jacobson L, Taylor A. The role of dual energy x-ray absorptiometry in aiding the diagnosis of pediatric osteogenesis imperfecta. Am J Orthop (Belle Mead NJ). 1998 Dec;27(12):797-801. PMID 9880097
- [Background] Roughley PJ, Rauch F, Glorieux FH. Osteogenesis imperfecta--clinical and molecular diversity. Eur Cell Mater. 2003 Jun 30;5:41-7; discussion 47. doi: 10.22203/ecm.v005a04. PMID 14562271
- [Background] Sillence DO, Senn A, Danks DM. Genetic heterogeneity in osteogenesis imperfecta. J Med Genet. 1979 Apr;16(2):101-16. doi: 10.1136/jmg.16.2.101. PMID 458828
- [Background] Maioli M, Gnoli M, Boarini M, Tremosini M, Zambrano A, Pedrini E, Mordenti M, Corsini S, D'Eufemia P, Versacci P, Celli M, Sangiorgi L. Genotype-phenotype correlation study in 364 osteogenesis imperfecta Italian patients. Eur J Hum Genet. 2019 Jul;27(7):1090-1100. doi: 10.1038/s41431-019-0373-x. Epub 2019 Mar 18. PMID 30886339
- [Background] Zionts LE, Nash JP, Rude R, Ross T, Stott NS. Bone mineral density in children with mild osteogenesis imperfecta. J Bone Joint Surg Br. 1995 Jan;77(1):143-7. PMID 7822373
- [Background] Hill CL, Baird WO, Walters SJ. Quality of life in children and adolescents with Osteogenesis Imperfecta: a qualitative interview based study. Health Qual Life Outcomes. 2014 Apr 16;12:54. doi: 10.1186/1477-7525-12-54. PMID 24742068
- [Background] Hald JD, Folkestad L, Harslof T, Brixen K, Langdahl B. Health-Related Quality of Life in Adults with Osteogenesis Imperfecta. Calcif Tissue Int. 2017 Nov;101(5):473-478. doi: 10.1007/s00223-017-0301-4. Epub 2017 Jul 4. PMID 28676897
- [Background] Vanz AP, van de Sande Lee J, Pinheiro B, Zambrano M, Brizola E, da Rocha NS, Schwartz IVD, de Souza Pires MM, Felix TM. Health-related quality of life of children and adolescents with osteogenesis imperfecta: a cross-sectional study using PedsQL. BMC Pediatr. 2018 Mar 2;18(1):95. doi: 10.1186/s12887-018-1077-z. PMID 29499676
- See also: Institutional webpage of Registries For Rare Hereditary Diseases — https://www.ior.it/en/curarsi-al-rizzoli/registries-rare-hereditary-diseases